CLINICAL TRIAL: NCT02608190
Title: Using Working Memory Training to Rehabilitate Unilateral Visual Neglect
Brief Title: Rehabilitating Unilateral Neglect Using Spatial Working Memory Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Principal Investigator, James Danckert, Professor, University of Waterloo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Danckert
Record Dates: First submitted 2015-11-11; First posted 2015-11-18 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hemispatial Neglect
MeSH Terms: conditions — Perceptual Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active training (Experimental): Patients will undergo active working memory training (see description of protocol).
  Interventions: Behavioral: Working memory training
- Passive training (Active Comparator): Patients will undergo passive working memory training (see description of protocol).
  Interventions: Behavioral: Working memory training

INTERVENTIONS:
Behavioral: Working memory training — See protocol

SUMMARY:
Purpose: Stroke is a common cause of death and disability in Canada. Injury to the right hemisphere of the brain and the parietal cortex in particular, is common and results in a disorder known as 'neglect' in 40% to 95% of patients. These patients fail to attend to or respond to events occurring in left space; the disorder is devastating for the patient and their caregivers with the patient becoming dependent on assistance for most activities of daily life (ADLs).

The project will implement two visual working memory (VWM) training programs to explore the influence of VWM training on neglect symptoms as well as activities of daily life.

Hypothesis: It is hypothesised that SWM training protocols will lead to improvements of neglect symptoms as well as improvement in ADLs.

The project will develop a novel rehabilitation strategy for treating the neglect syndrome.

Evidence from research in healthy participants employing video games to improve cognition along with research using working memory training protocols showing a broad range of benefits accruing to both trained and untrained tasks, suggests that the investigators approach has great potential to improve the core deficits of the neglect syndrome. Thus, WM training represents a promising avenue for rehabilitating neglect patients who demonstrate core deficits in both spatial attention and VWM to be highly interrelated functions.

DETAILED DESCRIPTION:
To examine the relationship between activities of daily living, attention and spatial working memory the investigators will have participants perform a range of clinical and experimental tasks over several sessions of testing. Below is an outline of the tasks to be used (attached are example of all tasks).

1. Clinical Tests: Neglect screenings: (a) The Behavioural Inattention Test (BIT) which includes pencil-and-paper or computer tablet tests of line bisection, figure copying and cancellation to assess for neglect. (b) The VRLAT as a more sensitive means to detect Neglect. Participants are asked to navigate through a virtual reality with a joystick. They are instructed to name objects presented on both sides of the virtual path while avoiding colliding with the objects along the way. The task takes approximately 5 minutes to complete. The Montreal Cognitive Assessment (MoCA): a brief screening tool for mild cognitive impairment
2. Spatial Attention Tasks: the covert orienting of visual attention task (COVAT), a computer task where participants fixate on a central point and detect targets presented at peripheral locations. Targets are preceded by peripheral cues that attract attention to one side or the other. Targets can appear at the cued location (i.e., a valid trial) or at the uncued location (i.e., an invalid trial). This task takes around 10 minutes to complete.
3. Visual Working Memory Task (VWM): One to three coloured squares arranged vertically in right space are presented for 500 ms in a computerized task. Following a delay a probe stimulus (bold rectangle) appears. Participants have to use the mouse to click on a colour bar to match the colour of the target that has previously occupied the highlighted space. This task takes about 30 minutes to complete.
4. Activities of daily living: The Frenchay Activities Index (FAI) is a short stroke specific questionnaire to assess functional status.

To assess the effects of working memory training on neglect two groups of neglect participants will be assigned to separate training protocols outlined below. Outcomes measures will include the tests outlined above and the VWM tasks themselves that were used in training.

1. Passive SWM training: the first group of participants will perform the VWM task described above, but do not actively engage in any specific component of the task (i.e., they passively respond to the stimuli appearing on the screen).
2. Active SWM training: the second training group will perform a task similar to the popular video game Guitar Hero. A sequence of virtual piano keys will be used on a tablet computer to simplify the game. Just as in Guitar Hero, a sequence of coloured targets, each corresponding to a specific piano key will gradually approach a target line at which point participants should hit the corresponding key of the virtual piano. A VWM component will be introduced to the task by presenting participants with a sequence of keys to touch followed by a brief delay. The investigators will manipulate load by changing the number of items in a given sequence (e.g., 1, 2, 3 and 5).

   After the delay participants will be required to repeat the sequence just presented by tapping the same keys on the tablet.
3. Training regimes and outcome measures: Two different lengths of training will be employed for both groups; 2 and 4 weeks, implemented as a between subjects factor. Participants will complete the training protocol for half an hour once per day using the tablet computer.

Outcome measures taken at 2 weeks, 4 weeks, 12 weeks include BIT, VRLAT COVAT, VWM, FAI.

Neglect participants will be contrasted to two control groups: healthy age-matched controls (recruited through WRAP) and a group of right brain damaged (RBD) participants without neglect.

ELIGIBILITY:
Inclusion Criteria:

* stroke presence of neglect symptoms

Exclusion Criteria:

* any other neurological or psychiatric syndrome
* any incapacity to perform the tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Improvement on behavioural tests | Measured at time zero (after intervention), 2 and 4 weeks post and 3 months post intervention.
  Performance on behavioural tests
Improvement on self-report measures | Measured at time zero (after intervention), 2 and 4 weeks post and 3 months post intervention.
  Changes to self-reported function in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: James Danckert, PhD, Principal Investigator — University of Waterloo
Locations (1):
- University of Waterloo, Waterloo, Ontario, Canada